CLINICAL TRIAL: NCT01129297
Title: Influence of the Glycemic and Ponderal Status on Tissues Gene Expression (Biological Tissue Collection)
Brief Title: A Biological Atlas of Severe Obesity (Biological Tissue Collection)
Acronym: ABOS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2006_0620; DGS 2006/0307 (Other: AFSSAPS)
Record Dates: First submitted 2010-05-04; First posted 2010-05-24 (Estimated); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Glucose Intolerance; Diabetes
Keywords: Obesity; surgery; genetic expression; collection of samples
MeSH Terms: conditions — Obesity; Glucose Intolerance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Liver samples before and at 1 and 5 years after bariatric surgery
  * Muscle samples before and at 1 year after bariatric surgery
  * Subcutaneous fat samples before and at 3 month and 1 year after bariatric surgery
  * Visceral fat samples in the great omentum before bariatric surgery
  * Intestinal samples during gastric by-pass surgery
  * Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- BMI ≥ 35 kg/m2 and diabetes: BMI (Body Mass Index) ≥ 35 kg/m2 and diabetes defined by a fasting blood glucose ≥ 7 mmol/l and/or ≥ to 11.1 mmol/l, 120 minutes after ingestion of glucose (oral glucose tolerance test)
- BMI ≥ 35 kg/m2 with intolerance glucose: BMI (Body Mass Index) ≥ 35 kg/m2 with intolerance glucose defined by a fasting blood glucose> 6 mmol/L and <7 mmol/l and / or> 7.8 mmol/l and <11.1 mmol/l , 120 minutes after ingestion of glucose (oral glucose tolerance test)
- BMI ≥ 35 kg/m2 without diabetes: BMI (Body Mass Index)≥ 35 kg/m2 without diabetes defined by a blood glucose ≤ 6 mmol/L and / or ≤ 7.8 mmol/l, 120 minutes after ingestion of glucose (oral glucose tolerance test)
- BMI <27 kg/m2 without diabetes: BMI (Body Mass Index) <27 kg/m2 without diabetes defined by a blood glucose ≤ 6 mmol/L and / or ≤ 7.8 mmol/l, 120 minutes after ingestion of glucose (oral glucose tolerance test)
- 27 < BMI < 35 kg/m2 without diabetes: BMI (Body Mass Index) <27 kg/m2 without diabetes defined by a blood glucose ≤ 6 mmol/L and / or ≤ 7.8 mmol/l, 120 minutes after ingestion of glucose (oral glucose tolerance test)

SUMMARY:
Type 2 diabetes and obesity are both multifactorial diseases resulting from gene-environment interactions. However, this interaction, as well as the specific effect of each polymorphism, remains poorly understood.

We now proposed a prospective cohort study to improve our understanding of the influence of phenotypic characteristics on gene expression in tissues involved in glucose and/or lipid metabolism by collecting different biological samples.

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) is a disease commonly associated with obesity, which is an important risk factor for this condition. More than 80% of the diabetic subjects are obese. By analogy with the metabolic syndrome, the close association between obesity and T2D justifies the recognition of a new disease entity named by the neologism "diabesity".

This study will examine the contribution of different genetic variants on "diabesity" development, by integrating multiple genomics approaches (linkage analysis on whole genome, transcriptomics and bioinformatics) and analysis of biological pathways in relevant animals models and humans.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Indication of abdominal surgery requiring a laparotomy or laparoscopy for bariatric surgery, cholecystectomy, or parietal surgical
* Phenotype corresponding to one of the following four cases :

  1. Body Mass Index ≥ 35 kg/m2 and diabetes defined by a fasting blood glucose ≥ 7 mmol/l and/or ≥ to 11.1 mmol/l, 120 minutes after ingestion of glucose (hyperglycemia caused by oral route)
  2. Body Mass Index ≥ 35 kg/m2 with intolerance glucose defined by a fasting blood glucose> 6 mmol/L and <7 mmol/l and/or> 7.8 mmol/l and <11.1 mmol/l , 120 minutes after ingestion of glucose (hyperglycemia caused by oral route)
  3. Body Mass Index ≥ 35 kg/m2 without diabetes defined by a blood glucose ≤ 6 mmol/L and / or ≤ 7.8 mmol/l, 120 minutes after ingestion of glucose (hyperglycemia caused by oral route)
  4. Body Mass Index <27 kg/m2 without diabetes defined by a blood glucose ≤ 6 mmol/L and / or ≤ 7.8 mmol/l, 120 minutes after ingestion of glucose (hyperglycemia caused by oral route)

5)27 <Body Mass Index <35 kg/m2 without diabetes defined by a blood glucose ≤ 6 mmol/L and / or ≤ 7.8 mmol/l, 120 minutes after ingestion of glucose (hyperglycemia caused by oral route)

Exclusion Criteria:

* unable to receive clear information
* refusal to sign the consent form
* pathology associated judged by the surgeon, may increase the risk of adverse events related to sampling tissue

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruiting: Clinical Medical Center from the north of France
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2006-06-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Study the influence of phenotypic characteristics on gene expression of tissues involved in glucose metabolism | Baseline
  Study the correlation between the glycemic status (fasting glucose and / or after ingestion of glucose) adjusted to the presence or absence of obesity (Body Mass Index) and gene expression in tissues involved in glucose metabolism before bariatric surgery

SECONDARY OUTCOMES:
Correlation between gene expression and tissue insulin resistance index (HOMA2) (The Homeostasis Model Assessment) | 1 year
  Insulin resistance is individually calculated by homeostasis model assessment(HOMA2) by determination of fasting glucose and insulin
Correlation between gene expression and tissue insulin resistance index (HOMA2) (The Homeostasis Model Assessment) | 2 years
  Insulin resistance is individually calculated by homeostasis model assessment(HOMA2) by determination of fasting glucose and insulin
Correlation between gene expression and tissue insulin resistance index (HOMA2) (The Homeostasis Model Assessment) | 5 years
  Insulin resistance is individually calculated by homeostasis model assessment(HOMA2) by determination of fasting glucose and insulin
Prospective assessment of clinical and biological features before and after bariatric surgery | 1 year
  Prospective assessment of clinical and biological features before and after bariatric surgery: weight, BMI, blood pressure, alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), prothrombin time, platelets, serum triglyceride, cholesterolemia, fasting blood glucose, fasting insulin, blood glucose and insulin 120 minutes after ingestion of glucose (oral glucose tolerance test)
Prospective assessment of clinical and biological features before and after bariatric surgery | 2 years
  Prospective assessment of clinical and biological features before and after bariatric surgery: weight, BMI, blood pressure, alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), prothrombin time, platelets, serum triglyceride, cholesterolemia, fasting blood glucose and fasting insulin, blood glucose and insulin 120 minutes after ingestion of glucose (oral glucose tolerance test)
Prospective assessment of clinical ans biological features before and after bariatric surgery | 5 years
  Prospective assessment of clinical and biological features before and after bariatric surgery: weight, BMI, blood pressure, alanine aminotransferase (ALT), gamma-glutamyl transferase (GGT), prothrombin time, platelets, serum triglyceride, cholesterolemia, fasting blood glucose and fasting insulin, blood glucose and insulin 120 minutes after ingestion of glucose (oral glucose tolerance test)
Genotype-Phenotype correlation | Baseline
  Genotype-Phenotype correlation based on medical and family history

CONTACTS AND LOCATIONS:
Overall Officials: Francois PATTOU, MD PhD, Principal Investigator — Lille University Hospital
Locations (1):
- Lille University Hospital, Lille, Nord, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lien F, Berthier A, Bouchaert E, Gheeraert C, Alexandre J, Porez G, Prawitt J, Dehondt H, Ploton M, Colin S, Lucas A, Patrice A, Pattou F, Diemer H, Van Dorsselaer A, Rachez C, Kamilic J, Groen AK, Staels B, Lefebvre P. Metformin interferes with bile acid homeostasis through AMPK-FXR crosstalk. J Clin Invest. 2014 Mar;124(3):1037-51. doi: 10.1172/JCI68815. Epub 2014 Feb 17. PMID 24531544
- [Derived] Raverdy V, Chatelain E, Lasailly G, Caiazzo R, Vandel J, Verkindt H, Marciniak C, Legendre B, Bauvin P, Oukhouya-Daoud N, Baud G, Chetboun M, Vantyghem MC, Gnemmi V, Leteurtre E, Staels B, Lefebvre P, Mathurin P, Marot G, Pattou F. Combining diabetes, sex, and menopause as meaningful clinical features associated with NASH and liver fibrosis in individuals with class II and III obesity: A retrospective cohort study. Obesity (Silver Spring). 2023 Dec;31(12):3066-3076. doi: 10.1002/oby.23904. PMID 37987186
- [Derived] Saux P, Bauvin P, Raverdy V, Teigny J, Verkindt H, Soumphonphakdy T, Debert M, Jacobs A, Jacobs D, Monpellier V, Lee PC, Lim CH, Andersson-Assarsson JC, Carlsson L, Svensson PA, Galtier F, Dezfoulian G, Moldovanu M, Andrieux S, Couster J, Lepage M, Lembo E, Verrastro O, Robert M, Salminen P, Mingrone G, Peterli R, Cohen RV, Zerrweck C, Nocca D, Le Roux CW, Caiazzo R, Preux P, Pattou F. Development and validation of an interpretable machine learning-based calculator for predicting 5-year weight trajectories after bariatric surgery: a multinational retrospective cohort SOPHIA study. Lancet Digit Health. 2023 Oct;5(10):e692-e702. doi: 10.1016/S2589-7500(23)00135-8. Epub 2023 Aug 29. PMID 37652841
- [Derived] Margerie D, Lefebvre P, Raverdy V, Schwahn U, Ruetten H, Larsen P, Duhamel A, Labreuche J, Thuillier D, Derudas B, Gheeraert C, Dehondt H, Dhalluin Q, Alexandre J, Caiazzo R, Nesslany P, Verkindt H, Pattou F, Staels B. Hepatic transcriptomic signatures of statin treatment are associated with impaired glucose homeostasis in severely obese patients. BMC Med Genomics. 2019 Jun 3;12(1):80. doi: 10.1186/s12920-019-0536-1. PMID 31159817